CLINICAL TRIAL: NCT06387368
Title: Prospective, Multicenter, Randomized, Parallel Controlled Clinical Study on the Efficacy and Safety of Huaier Granules Combined With Capecitabine Versus Capecitabine Alone in the Treatment of Unresectable Pancreatic Cancer
Brief Title: Clinical Study of Huaier Granule in the Treatment of Unresectable Pancreatic Cancer
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Xi'an Jiaotong University (Other)
Collaborators: LinkDoc Technology (Beijing) Co. Ltd. (Industry); Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Zheng Wang, professor, Xi'an Jiaotong University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HE-202303
Record Dates: First submitted 2024-04-23; First posted 2024-04-29 (Actual); Last update posted 2024-04-29 (Actual); Status verified 2024-04

CONDITIONS: Pancreatic Cancer Non-resectable
Keywords: Huaier Granules; Capecitabine; Unresectable Pancreatic Cancer; Efficacy and Safety
MeSH Terms: interventions — Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Huaier treatment group (Experimental): The subjects received a combination of Huaier granules and capecitabine regimen.The subject takes Huaier granules orally, 10g once, three times a day; take capecitabine 1250mg/m^2 orally , twice a day (2500mg/m^2/d), day 1-14, once every 3 weeks.
  Interventions: Drug: Huaier Granule
- Control group (Active Comparator): The subjects received the capecitabine monotherapy regimen. The subjects take capecitabine orally, 1250mg/m^2, twice a day (2500mg/m^2/d), day for 1-14 days, once every 3 weeks.
  Interventions: Drug: Capecitabine

INTERVENTIONS:
Drug: Huaier Granule — Huaier Granules: Oral administration, 10g once, 3 times a day. Capecitabine: oral administration, 1250mg/m^2, twice a day (2500mg/m^2/d), day 1-14, once every 3 weeks.
  Other Names: Z20000109#NMPA Approval Number#
  Arms: Huaier treatment group
Drug: Capecitabine — Oral administration, 1250mg/m^2, twice a day (2500mg/m^2/d), day 1-14, once every 3 weeks.
  Other Names: Standard chemotherapy
  Arms: Control group

SUMMARY:
This is a prospective, multicenter, randomized, open, parallel controlled clinical study to evaluate the efficacy and safety of Huaier Granules combined with capecitabine in the treatment of unresectable pancreatic cancer.

DETAILED DESCRIPTION:
This study is a prospective, multicenter, randomized, open label, parallel controlled clinical study. It is expected to include approximately 488 patients diagnosed with unresectable pancreatic adenocarcinoma by tissue or cellular pathology who visited the selected research center from April 2024 to March 2026. The treatment regimen will be capecitabine monotherapy orally. Among them, the Huaier group uses "capecitabine+Huaier granules", and is expected to include 244 cases; The control group received capecitabine and is expected to include 244 cases.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old, regardless of gender.
* The patient has a clear evaluable lesion (RECIST 1.1) and is diagnosed with pancreatic adenocarcinoma through tissue or cellular pathology. Clinical evaluation suggests that radical surgical resection cannot be performed (due to jaundice and gastrointestinal obstruction caused by tumor compression, stent treatment or normal inclusion of biliary and gastrointestinal anastomosis can be performed).
* Patients voluntarily give up conversion therapy, local radiation therapy, targeted immunity, and other programs.
* The patient voluntarily choose chemotherapy, and the plan is to take capecitabine monotherapy orally.
* ECOG score 0-3 points.
* The patients voluntarily participate in and cooperates with all aspects of the research, including but not limited to cooperating with treatment and follow-up, cooperating with the researcher in data collection, not actively taking other treatments, and signing a written informed consent form.

Exclusion Criteria:

* Known to be allergic to the components of Huaier granules or to avoid or use Huaier granules with caution (Huaier group).
* Patients with difficulty swallowing, complete or incomplete gastrointestinal obstruction (excluding those who have undergone gastrointestinal stenting or diversion surgery due to tumor related gastrointestinal obstruction and have a normal diet, can be included in the study normally), active gastrointestinal bleeding, perforation, and other oral medication difficulties.
* After actively reducing jaundice (including but not limited to bile duct/gallbladder puncture external drainage, nasobiliary duct external drainage, biliary stent internal drainage, biliary intestinal anastomosis internal drainage, etc.), the levels of aspartate aminotransferase, alanine aminotransferase, or total bilirubin are still 2.5 times higher than the upper limit of normal values.
* History of merging with other malignant tumors.
* Patients with concomitant myocardial infarction, cerebral infarction, and other thromboembolic diseases requiring surgical treatment.
* Concomitant severe infection.
* Child-Pugh C-grade liver function, renal function 2-5 grades (glomerular filtration rate<90ml/min).
* Pregnant or lactating women or those planning to conceive.
* The patient has received other traditional Chinese patent medicines and simple preparations with anti-tumor effect, chemotherapy or physical therapy in the past 4 weeks(including but not limited to compound cantharidin capsules, cinobufotalin capsules, Kangai injection, please refer to the drug instructions for details).
* Suffering from serious mental illness or other reasons that the researcher deems unsuitable to participate in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 488 (Estimated)
Dates: Start 2024-05 (Estimated); Primary Completion 2028-03 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Overall survival | Start of treatment until 2-year follow-up
  It is defined as the time from the day of patient randomization to death due to any reason.

SECONDARY OUTCOMES:
Objective response rate | Start of treatment until 2-year follow-up
  It is defined as the proportion of patients whose tumors have shrunk to a certain amount and maintained for a certain period of time, generally understood as the sum of CR and PR(CR ,complete remission ,all target lesions disappear, maintained for 4 weeks; PR ,partial remission ,it is defined as a reduction of at least 30% in the sum of the longest diameters of the target lesion compared to baseline, maintained for 4 weeks).
Progression free survival | Start of treatment until 2-year follow-up
  It is defined as the period between the start of treatment and the observation of disease progression or death due to any reason for patients with pancreatic cancer in this study.
Conversion surgery rate | Start of treatment until 2-year follow-up
  It is defined as the proportion of patients diagnosed as locally advanced pancreatic cancer before surgery (stage III) who can accept radical surgery after clinical evaluation; The proportion of patients with oligometastatic lesions (belonging to stage IV) who have no new lesions and significant regression of the metastatic lesions after treatment, and whose primary lesions can be removed (regardless of whether they can be removed before treatment) are clinically assessed as eligible for radical surgery.
The incidence and severity of adverse events (AE) and severe adverse events (SAE) | Start of treatment until 2-year follow-up
  The definitions and severity grading of AE and SAE refer to the corresponding descriptions in the definition and evaluation section of AE. The incidence rate is defined as the proportion of patients with AE and SAE to the corresponding total population.
The incidence and severity of ADR, severe adverse reactions (SADR), suspicious and unexpected severe adverse reactions (SUSAR) | Start of treatment until 2-year follow-up
  The definitions and severity grading of ADR, severe ADR, and SUSAR refer to the corresponding descriptions in the definition and evaluation section of AE. The incidence rate is defined as the proportion of patients with ADR, severe ADR, and SUSAR to the corresponding total population.

CONTACTS AND LOCATIONS:
Overall Officials: Zheng Wang, PhD, Principal Investigator — First Affiliated Hospital Xi'an Jiaotong University